CLINICAL TRIAL: NCT05523258
Title: The Effect and Mechanism of Computerized Cognition Training on the Incidence of Postoperative Cognitive Dysfunction After Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mu Dong Liang (Other)
Responsible Party: Sponsor-Investigator, Mu Dong Liang, Deputy chief physician, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-156
Record Dates: First submitted 2022-08-28; First posted 2022-08-31 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Cognitive Dysfunction(POCD)
Keywords: POCD; cardiac surgery; cognitive training
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in this group will receive computerized cognition training, including processing speed, attention, perception, long-term memory, working memory, calculation, executive control, reasoning and problem solving. The training program and its difficulty are constantly adjusted with the patients' training performance.
  Interventions: Behavioral: Computerized cognition training
- Control group (Sham Comparator): Patients in this group will receive basic training based on tablet computer, and the subjects will receive five training tasks of processing speed and attention, which are fixed in difficulty and scheme. The training methods and intensity are similar to the intervention group.
  Interventions: Behavioral: Basic training based on tablet computer

INTERVENTIONS:
Behavioral: Computerized cognition training — The researchers distribute tablet computers for the patients. The patients in this group receive cognitive function training under the guidance of a full-time cognitive function trainer. The training time is about 45-60 minutes every time, and the frequency is twice a day until the operation. After the operation, cognitive function training should be started as soon as possible when the patient meets the following conditions including Glasgow score ≥ 12, no mechanical ventilation and no sedative drugs. The training intensity is the same as that before operation, generally starting from the 2nd to 3rd day after operation and continuing to discharge or the 7th day after operation.
  Arms: Intervention Group
Behavioral: Basic training based on tablet computer — The researchers distribute the same tablet computer to the patients. The patients in this group receive basic training under the guidance of a full-time cognitive function trainer. The training duration is the same as that of the test group.
  Arms: Control group

SUMMARY:
Whether enough time and high-quality cognitive training will reduce the incidence of postoperative cognitive dysfunction after cardiac surgery.

DETAILED DESCRIPTION:
Firstly, after patients are admitted, the researchers will visit every patient, introduce the study protocol, the risks and rights of the subjects to them in detail, and obtain their signed informed consent. Then, researches will collect the baseline data of the patients and complete the baseline status data measurement, including cognitive function, sleep quality, anxiety and depression scores, multi-channel EEG recorder monitoring and functional magnetic resonance examination.

According to the results of randomization, the intervention will be carried out according to the study protocol.

The day before the operation, EEG cortical network connection status, cognitive function, sleep quality, anxiety and depression scores will be measured after the intervention to understand the effect of preoperative intervention on brain function.

On the day of operation, anesthesia and operation will be performed according to clinical routine. And the multi-channel EEG will be detected after induction of anesthesia and during the period of sedation and recovery.When the patient meets the appropriate conditions, cognitive function training will be started as soon as possible.

Researches will evaluate the patients' sleep quality and the incidence of delirium in the first six days after the operation. They will also evaluate cognitive function, sleep quality, anxiety and depression scores, and conduct postoperative delirium evaluation, multi-channel EEG recorder monitoring, functional magnetic resonance examination on the seventh day after operation.The cognitive function, sleep quality, anxiety and depression scores will be measured 30 days after operation.

The Clinical Research Institute of Peking University undertakes the work of data collection and analysis of this project. A electronic data acquisition system based on network is used for data acquisition, where researchers need to input the research data accurately, timely and comprehensively. The audit and quality control will be fed back to the researchers in time. The researchers need to check the feedback one by one and record the check results in detail.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in this study voluntarily;
* Age ≥ 60 years old；
* Patients who intend to accept elective coronary artery bypass grafting or valve replacement；
* The preoperative hospital stay is expected to be 5 days or more.

Exclusion Criteria:

* Definite diagnosis of senile dementia and Montreal Cognitive Assessment(MoCA) score ≤ 18;
* Patients with severe visual or hearing impairment who cannot complete the cognitive function assessment;
* Patients with limb movement disorder who cannot complete the cognitive function assessment;
* Patients with claustrophobia who cannot complete functional magnetic resonance imaging(fMRI) examination;
* The expected survival time is less than 1 month;
* Patients within 3 months or participating in other clinical trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative 7-day cognitive dysfunction | The 7th day after operation

SECONDARY OUTCOMES:
Postoperative 7-day changes of cognitive scores | The 7th day after operation
Postoperative 7-day changes of cortical network connectivity function | The 7th day after operation
Postoperative 7-day changes of sleep quality | The 7th day after operation
Incidence of postoperative delirium within 7 days | Within 7 days after operation
Incidence of postoperative 30-day cognitive dysfunction | The 30th day after operation
Postoperative 30-day main complications and mortality | The 30th day after operation